CLINICAL TRIAL: NCT04228536
Title: Chronic Pain After Groin Hernia Surgery in Women
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Region Jämtland Härjedalen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00041
Record Dates: First submitted 2019-08-13; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-02

CONDITIONS: Hernia, Inguinal; Hernia, Femoral
Keywords: chronic pain
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Femoral; Chronic Pain | interventions — tetraethylpyrazine; Wound Healing; tetra-4-amidinophenoxypropane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Totally ExtraPeritoneal (TEP) repair
Procedure: TransAbdominal PrePeritoneal (TAPP) repair
Procedure: Open anterior mesh repair (OAM)
  Other Names: Lichtenstein
Procedure: Combined Anterior and Posterior technique (CAP)
  Other Names: Plug; Prolene Hernis System (PHS); Onstep; TransInguinalPrePeritoneal repair (TIPP)
Procedure: Open PrePeritoneal Mesh technique (OPPM)
  Other Names: Nyhus; Stoppa; Hives
Procedure: Sutured Repair
  Other Names: McVay; Bassini; Shouldice; Marcy

SUMMARY:
The goal of this study was to evaluate chronic pain and reoperation rates due to recurrence after groin hernia surgery in women compared to men and surgical method.

DETAILED DESCRIPTION:
INTRODUCTION:

Groin hernia surgery in women is much less common than in men, still women represent a large patient group since groin hernia surgery is one of the most common operations in general surgery. In Sweden, approximately 16 000 groin hernia surgeries are being performed annually, of these 8 % are performed in women. Management and method of repair in women is largely based on subgroup analyses and register studies, there is a lack of randomised controlled trials focusing on women. Previous studies have shown that femoral hernias are more common in women than in men, that women have a higher risk of emergency operation, and a higher incidence of reoperation which serves as a marker of recurrence. Chronic pain is common after herniorraphy and an important quality marker of the performed surgery. There are indications that women suffer of higher rates of both short term and chronic post-herniorraphy pain. The introduction of mesh techniques in groin hernia surgery has considerably decreased recurrence rates. To further improve outcome after groin hernia surgery in women there is a need for more evidence of the most appropriate surgical approach in terms of chronic pain.The goal of this study was to evaluate chronic pain and reoperation rates due to recurrence after groin hernia surgery in women compared to men.

METHODS

This study is based on a patient reported outcome measure (PROM) questionnaire, crosslinked to the Swedish Hernia Registry one year after primary surgery. What the investigators would like to call a Register-PROM-study.

The Swedish Hernia Registry (SHR)

SHR is a nationwide registry which covers more than 95% of all performed groin hernia repairs in Sweden. Patients are included upon surgery. Registered parameters include details about hernia anatomy, method of repair, American Society of Anesthesiologists (ASA) Physical Status and early complications (within 30 days), among others. Using the Swedish personal identity number, where each inhabitant has a unique number, it is possible to follow patients regardless of where the participants have their primary or recurrence operation.

Questionnaire

To measure the postoperative pain one year after primary operation a shortened version of the previously validated Inguinal Pain Questionnaire (IPQ) was used. Patients were asked to grade the worst pain the participants had felt in the operated groin during the last week. Scores were:

1. No pain.
2. Pain present, but easily ignored.
3. Pain present, cannot be ignored, but does not interfere with everyday activities.
4. Pain present, cannot be ignored, and interferes with concentration on everyday activities.
5. Pain present, interferes with most activities.
6. Pain present, necessitating bed rest.
7. Pain present, prompt medical advice sought. Scores of 1-3 were defined as no pain and scores of 4-7 as chronic pain.

Data Collection

The questionnaire is sent by regular mail to everyone included in the SHR one year after surgery. Answers are recorded in the SHR. The participants are able to answer the questionnaire by mail or a web based questionnaire. Postal addresses were obtained through the Swedish population register. If no response had been received within 1 month a reminder was sent. A previous study with a similar cohort has analyzed loss to follow up and reliability of the method.

ELIGIBILITY:
Inclusion Criteria:

* All patients 15 years and older included in the SHR between 1 Sept. 2012 and 31 Aug 2017. Both elective and acute surgery is included.

Exclusion Criteria:

* Patients not responding to questionnaire. Patients were the first operation during inclusion period was a reoperation.
* Patient with bilateral operations during the study-period are only included once.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients 15 years and older included in the SHR between 1 Sept. 2012 and 31 Aug 2017.
Sampling Method: Probability Sample
Enrollment: 44915 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of chronic pain in women 1 year after groin hernia surgery. | 1 year after groin hernia surgery
  Using Inguinal Pain Questionnaire (IPQ) for patient reported outcome measure.
Rate of chronic pain in men 1 year after groin hernia surgery. | 1 year after groin hernia surgery
  Using Inguinal Pain Questionnaire (IPQ) for patient reported outcome measure.

SECONDARY OUTCOMES:
Rate of reoperation for recurrence. | Through study completion, minimum follow up 1 year

OTHER OUTCOMES:
Age as a risk factors for chronic pain after groin hernia surgery | 1 year after groin hernia surgery
  Using Inguinal Pain Questionnaire (IPQ) for patient reported outcome measure.
Sex as a risk factors for chronic pain after groin hernia surgery | 1 year after groin hernia surgery
  Using Inguinal Pain Questionnaire (IPQ) for patient reported outcome measure
Hernia anatomy as a risk factors for chronic pain after groin hernia surgery | 1 year after groin hernia surgery
  Using Inguinal Pain Questionnaire (IPQ) for patient reported outcome measure
Method of repair as a risk factors for chronic pain after groin hernia surgery | 1 year after groin hernia surgery
  Using Inguinal Pain Questionnaire (IPQ) for patient reported outcome measure
Acute surgery as a risk factors for chronic pain after groin hernia surgery | 1 year after groin hernia surgery
  Using Inguinal Pain Questionnaire (IPQ) for patient reported outcome measure
Annual surgeon volume as a risk factors for chronic pain after groin hernia surgery | 1 year after groin hernia surgery
  Using Inguinal Pain Questionnaire (IPQ) for patient reported outcome measure.
ASA grade as a risk factors for chronic pain after groin hernia surgery | 1 year after groin hernia surgery
  The ASA physical status classification system is a system for assessing the fitness of patients before surgery.
BMI as a risk factors for chronic pain after groin hernia surgery | 1 year after groin hernia surgery
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Pär Nordin, M.D., Ph.D., Principal Investigator — Umeå University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Franneby U, Gunnarsson U, Andersson M, Heuman R, Nordin P, Nyren O, Sandblom G. Validation of an Inguinal Pain Questionnaire for assessment of chronic pain after groin hernia repair. Br J Surg. 2008 Apr;95(4):488-93. doi: 10.1002/bjs.6014. PMID 18161900
- [Derived] Jakobsson E, Lundstrom KJ, Holmberg H, de la Croix H, Nordin P. Chronic Pain After Groin Hernia Surgery in Women: A Patient-reported Outcome Study Based on Data From the Swedish Hernia Register. Ann Surg. 2022 Feb 1;275(2):213-219. doi: 10.1097/SLA.0000000000005194. PMID 35007224